CLINICAL TRIAL: NCT04952519
Title: Efficacy of Amantadine Treatment in COVID-19 Patients
Acronym: TITAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The annual analysis did not show the efficacy of the investigational medicinal product in this application, therefore the study was not continued.
Sponsor: Noblewell (Industry)
Collaborators: Medical Research Agency, Poland (Other Government); Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00980.045; 2021-000981-13 (EudraCT Number)
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2021-07

CONDITIONS: Patients With Moderate or Severe COVID-19
Keywords: SARS-COV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amantadine (Experimental)
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Patients are treated with high doses of amantadine.

SUMMARY:
Demonstration of the efficacy of amantadine over placebo in the population of patients with moderate or severe COVID-19 in the initial stage of the disease treated in the hospital

DETAILED DESCRIPTION:
Use of high-doses of amantadine in hospitalized patients in the early phase of moderate or severe COVID-19, compared to placebo, will shorten the duration of the disease and reduce the risk of death and treatment with invasive mechanical ventilation in Intensive Care Units (ICU).

ELIGIBILITY:
Inclusion Criteria:

1. Age of respondents - 18 years and older.
2. Confirmation of SARS-CoV-2 infection by PCR
3. Hospitalized patient with COVID-19, defined according to the following criteria (all of the following criteria must be present):

   1. radiological (X-ray of klp or TK klp) features of pneumonia,
   2. blood saturation (SaO2) measured at rest in the absence of oxygen <95%,
   3. it is not necessary to apply on the day of patient enrollment: high-flow oxygen therapy or mechanical ventilation (non-invasive or invasive).
4. Time up to 10 days from the onset of COVID-19 symptoms. The onset of COVID-19 symptoms is the first day on which the first symptom typical for SARS-CoV-2 or COVID-19 infection (in the opinion of the attending physician at the center) occurred, such as: fever, cough, shortness of breath, changes in taste or smell , muscle pain, chest pain, diarrhea, nausea, vomiting, sore throat, nasal congestion.

Exclusion Criteria:

1. Pregnancy or lactation
2. Presence of medical contraindications for inclusion in the examination in the opinion of the attending physician, in particular:

   a) comorbidities: i) clinically significant hepatic or renal insufficiency; ii) epilepsy or seizures (current or history of); iii) psychiatric or somatic diseases (present or in a history of agitation or confusion, delirium syndromes or exogenous psychoses); iv) cardiovascular diseases such as: severe congestive heart failure, cardiomyopathy, myocarditis, grade II-IV AV block, bradycardia, QT prolongation, perceived U waves or family history of congenital long QT syndrome, severe ventricular arrhythmias a history of heart (including torsade de pointes); v) diseases or conditions that significantly reduce the immunity of a patient (e.g. solid organ transplant, bone marrow transplantation (BMT), AIDS, immune biologics and / or high-dose steroids (> 20 mg prednisone daily).

   b) hypersensitivity to any component of the preparation, c) parallel use of drugs that prolong the QT interval, d) hypokalemia or hypomagnesaemia, e) untreated angle-closure glaucoma, f) use of amantadine currently or in the last 3 months prior to study inclusion; g) participation in another clinical program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Time to recovery | 28 days
  Time to recovery, defined as the first day during the 28-day clinical follow-up during which the patient's clinical condition is graded 1, 2, or 3 on an eight-point "Normal Symptom Score"

CONTACTS AND LOCATIONS:
Overall Officials: Adam Barczyk, Prof., Study Director — Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice
Locations (12):
- Poland (12):
  - I Klinika Chorób Płuc i Gruźlicy z Pododdziałem Chemioterapii - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Szpital Tymczasowy Zespół Opieki Zdrowotnej, Bolesławiec
  - Oddział Chorób Płuc i Niewydolności Oddychania z Pododdziałem NWM i Pododdziałem Zaburzeń Oddychania w Czasie Snu, Kujawsko - Pomorskie Centrum Pulmonologii w Bydgoszczy, Bydgoszcz
  - Oddział Chorób Płuc i Chemioterapii - Szpital Powiatowy w Chrzanowie, Chrzanów
  - Oddział Pneumonologii Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Oddział Pulmonologii Szpital Powiatowy w Limanowej Imienia Miłosierdzia Bożego, Limanowa
  - Oddział Pulmonologiczny Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Szpital Tymczasowy w Pyrzowicach, Pyrzowice
  - Oddział Chorób Płuc; Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Oddział gruźlicy i chorób płuc; Lubuski Szpital Specjalistyczny Pulmonologiczno-Kardiologiczny w Torzymiu Spółka z o.o., Torzym
  - Klinika Alergologii, Chorób Płuc i Chorób Wewnętrznych, Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Tymczasowy Szpital Narodowy, CSK MSWiA, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barczyk A, Czajkowska-Malinowska M, Farnik M, Barczyk M, Boda L, Cofta S, Dulawa J, Dyrbus M, Harat R, Huk M, Kotecka S, Nahorecki A, Nasilowski J, Naumnik W, Przybylski G, Slabon-Willand M, Skoczynski S, Wita K, Ziolo G, Kuna P. Efficacy of oral amantadine among patients hospitalised with COVID-19: A randomised, double-blind, placebo-controlled, multicentre study. Respir Med. 2023 Jun;212:107198. doi: 10.1016/j.rmed.2023.107198. Epub 2023 Mar 15. PMID 36931576